CLINICAL TRIAL: NCT07377279
Title: Acupuncture and Compression for the Prevention of Peripheral Neuropathy Induced by Taxane-based Chemotherapy in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: Acupuncture and Compression for the Prevention of CIPN in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYSKY-2025-870-02
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy (CIPN)
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compression (Experimental): Latex gloves and compression stockings are worn during chemotherapy.
  Interventions: Other: Compression
- Acupuncture (Experimental): Electroacupuncture treatment is administered after each chemotherapy cycle and continuing consecutively for 3-5 days.
  Interventions: Other: Acupuncture
- Compression combined with acupuncture (Experimental): Compression therapy will be administered during chemotherapy, combined with consecutive electroacupuncture for 3-5 days after each chemotherapy cycle.
  Interventions: Other: Compression combined with acupuncture
- Sham acupuncture (Placebo Comparator): A shallow needling at non-acupoint sites (sham acupuncture) is inserted superficially to a depth of 2-3 mm without manipulation.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Compression — Two layers of latex gloves are worn on both hands, and Class II compression stockings are worn on both feet. The devices are donned 30 minutes before chemotherapy initiation and removed 30 minutes after chemotherapy completion.
  Arms: Compression
Other: Acupuncture — Acupuncture is administered consecutively for 3-5 days starting from Day 1 post each chemotherapy cycle, with electrical stimulation applied for 20-30 minutes per session. The selected acupoints included: PC6, LI4, SI3, ST36, SP6, LR3, SP4, EX-LE10.
  Arms: Acupuncture
Other: Sham acupuncture — A shallow needling at non-acupoint sites (sham acupuncture) is adopted. The stimulation locations are non-acupoint areas 1-2 cun away from the standard acupoint positions. For the sham acupuncture group, needles are inserted superficially to a depth of 2-3 mm without manipulation, with the endpoint of no deqi sensation. Operational elements including needle type, patient posture, disinfection method, needle insertion technique, needle retention time, and needle withdrawal technique are identical between the sham acupuncture group and the active acupuncture group.
  Arms: Sham acupuncture
Other: Compression combined with acupuncture — Two layers of latex gloves are worn on both hands, and Class II compression stockings are worn on both feet. The devices are donned 30 minutes before chemotherapy initiation and removed 30 minutes after chemotherapy completion. Acupuncture is administered consecutively for 3-5 days starting from Day 1 post each chemotherapy cycle, with electrical stimulation applied for 20-30 minutes per session. The selected acupoints included: PC6, LI4, SI3, ST36, SP6, LR3, SP4, EX-LE10.
  Arms: Compression combined with acupuncture

SUMMARY:
As a core component of comprehensive breast cancer treatment, chemotherapy frequently induces chemotherapy-induced peripheral neuropathy (CIPN), particularly with taxane-based agents. The incidence of CIPN reaches 68.1% within the first month of chemotherapy, and over 30% of patients experience persistent symptoms for more than 6 months. The resulting sensorimotor dysfunction significantly impairs patients' quality of life, necessitates dose reduction or treatment discontinuation, and ultimately affects survival outcomes. Currently, no prophylactic pharmacological or non-pharmacological interventions have received Grade I recommendations in domestic or international guidelines and expert consensuses. The compression therapy demonstrated definite preventive value in the POLAR trial. Its low cost and high tolerability confer substantial clinical applicability, earning it a Grade III recommendation in ESMO guidelines. Meanwhile, single-arm trials of acupuncture have reported a 51.2% symptom relief rate and a trend toward reduced high-grade CIPN. As non-pharmacological interventions, acupuncture and compression therapy hold complementary potential in preventing taxane-induced CIPN: compression therapy locally blocks drug exposure, while acupuncture systemically regulates neural function.However, three core challenges persist in the current research field: insufficient evidence quality for single-intervention strategies, lack of systematic evaluation of combined interventions, and the absence of risk-stratified prevention models. To address these gaps, this study aims to conduct a prospective randomized controlled trial to concurrently evaluate the preventive efficacy of compression therapy, acupuncture, and their combination for taxane-induced CIPN. The goal is to provide high-level evidence-based medicine to support the development of individualized prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old and have signed an informed consent form;
2. Patients with histologically confirmed non-recurrent early or intermediate-stage breast cancer;
3. Patients scheduled to receive cyclical adjuvant or neoadjuvant chemotherapy based on taxane drugs (4-cycle or single-cycle regimen);
4. No prior exposure to breast cancer-related chemotherapy, immunotherapy, or endocrine therapy;
5. Cardiac echocardiography showing cardiac ejection fraction within normal range;
6. Eastern Cooperative Oncology Group (ECOG) physical status ≤1;
7. No psychiatric or cognitive impairments, capable of understanding and completing assessment scales;
8. No CIPN at baseline (NCI-CTCAE 5.0 and TNSc grading ≤0);
9. Good organ function meeting the following criteria: Hb ≥90g/L, WBC ≥3.5×10⁹/L, platelets ≥100×10⁹/L, neutrophils ≥1.5×10⁹/L, AST ≤3× upper limit of normal, ALT ≤3× upper limit of normal, bilirubin ≤1.5× upper limit of normal, serum creatinine ≤1.5× upper limit of normal;
10. Fertile women must agree to use effective contraception for 7 days before first dosing through 24 weeks post-treatment. Fertile women must have a negative serum pregnancy test within 7 days before first dosing.

Exclusion Criteria:

1. Patients with active infections, skin lesions on hands/feet, or contraindications to chemotherapy, acupuncture, or compression therapy;
2. Patients with prior exposure to neurotoxic agents (e.g., taxanes, oxaliplatin, platinum-based drugs, vincristine) or platinum-containing chemotherapy regimens;
3. Patients who received acupuncture for other conditions within the past month;
4. Patients with conditions predisposing to peripheral neuropathy symptoms (e.g., alcoholism, uremia, diabetes, autoimmune disorders, rheumatoid arthritis, cervical spondylosis, severe mental illness, severe trauma);
5. Patients with Raynaud's syndrome, cold intolerance, peripheral arterial ischemia, or hand-foot syndrome;
6. Patients receiving medications that may mask CIPN symptoms (e.g., SSNRI, SSRI, tricyclic antidepressants, B-complex vitamins);
7. Patients with lymphedema in acupuncture stimulation areas;
8. Patients with phobia of electroacupuncture or stainless steel needle allergy;
9. Patients with severe non-malignant conditions that may compromise treatment adherence or pose risks;
10. Patients undergoing concurrent anti-tumor therapy or clinical trials;
11. Patients with dementia, cognitive impairment, or psychiatric conditions affecting informed consent comprehension;
12. Patients with known allergy history or contraindications to trial procedures;
13. Patients with uncontrolled cardiac symptoms or conditions, including: (1) NYHA class 2 or higher heart failure; (2) unstable angina; (3) myocardial infarction within the past year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment;
14. Cardiac pacemaker implantation;
15. Known hereditary or acquired bleeding/thrombosis predispositions (e.g., hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥2 CIPN at 12 weeks after the initiation of chemotherapy | 12 weeks after the initiation of chemotherapy
  The incidence of CIPN ≥ grade 2 is assessed according to the NCI-CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Incidence of CIPN | 6 and 12 weeks after chemotherapy initiation, 12 and 24 weeks after chemotherapy completion
  The incidence of CIPN at 6 and 12 weeks after chemotherapy initiation, and at 12 and 24 weeks after chemotherapy completion
Incidence of grade ≥2 CIPN at 6 weeks after chemotherapy initiation, 12 and 24 weeks after chemotherapy completion | 6 weeks after chemotherapy initiation, 12 and 24 weeks after chemotherapy completion
  The incidence of CIPN ≥2 grade at 6 weeks after chemotherapy initiation, 12 weeks after chemotherapy completion, and 24 weeks after chemotherapy completion.
Assessment of quality of life via the EORTC QLQ-C30 questionnaire. | Every 6 weeks until the end of chemotherapy; 12 and 24 weeks after the end of chemotherapy.
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30). It contains 30 items and measures 5 functional scales (physical, role, emotional, cognitive, and social), a global health and quality of life scale, 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact). The global health and quality of life scale uses a 7-point scale scoring with anchors (1=very poor and 7=excellent); the other items are scored on a 4 point scale (1=not at all, 2=a little, 3= quite a bit, 4=very much).
Assessment of sensation and motor function via the EORTC QLQ-CIPN20 questionnaire. | Every 6 weeks until the end of chemotherapy; 12 and 24 weeks after the end of chemotherapy.
  Patient reported outcomes via the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale (EORTC QLQ-CIPN20). It contains 20 items divided into 3 subscales assessing sensory, motor and autonomic symptoms. Each item is scored on a Likert scale ranging from 1 'not at all' to 4 'very much'. Scores are transformed to a 0-100 scale, with higher scores representing more complaints.
Nail toxicity | Every 6 weeks until the end of chemotherapy; 12 and 24 weeks after the end of chemotherapy.
  Nail toxicity is assessed according to the National Cancer Institute Toxicity Criteria 4.0 (NCI 4.0).
Objective neurological function | Every 6 weeks until the end of chemotherapy; 12 and 24 weeks after the end of chemotherapy.
  Use quantitative sensory testing to assess vibration perception (128Hz tuning fork, dorsal threshold>8 seconds) and tactile sensation (10g monofilament, no response at ≥2 of 4 hand/foot points).
Adverse event incidence rate | 8 months (during taxane therapy and follow up).
  Adverse events at all levels associated with treatment and interventions

OTHER OUTCOMES:
Blood sample analysis | 3 months (before and after taxane therapy)
  Compare the differences in NfL levels, metabolites and other aspects among blood samples from different groups to identify molecular markers potentially associated with the occurrence of CIPN.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Tumor Center, Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China